CLINICAL TRIAL: NCT02313883
Title: A Phase I/II Study to Evaluate the Safety, Tolerability and Efficacy of PerioSept® and Scaling and Root Planing in Subjects With Periodontitis
Brief Title: A Phase I/II Study to Evaluate the Safety and Efficacy of PerioSept® as Adjunct to SRP in Subjects With Periodontitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Geistlich Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PSPD 1-2
Record Dates: First submitted 2014-12-08; First posted 2014-12-10 (Estimated); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Periodontitis
Keywords: periodontitis; taurolidine (PerioSept(r)); scaling and root planing
MeSH Terms: conditions — Periodontitis | interventions — taurolidine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- SRP only (Placebo Comparator): Scaling and root planing only
  Interventions: Drug: PerioSept(r)
- SRP and Placebo (Placebo Comparator): Scaling and root planing followed by placebo drug administration
  Interventions: Drug: PerioSept(r)
- SRP and 0.3% PerioSept(r) (Experimental): Scaling and root planing followed by 0.3% PerioSept(r) drug administration
  Interventions: Drug: PerioSept(r)
- SRP and 1 % PerioSept(r) (Experimental): Scaling and root planing followed by 1% PerioSept(r) drug administration
  Interventions: Drug: PerioSept(r)
- SRP and 3% PerioSept(r) (Experimental): Scaling and root planing followed by 3% PerioSept(r) drug administration
  Interventions: Drug: PerioSept(r)

INTERVENTIONS:
Drug: PerioSept(r) — Taurolidine is derived from the amino acid taurine and has antimicrobial and immune modulating properties
  Other Names: Taurolidine

SUMMARY:
A Pharmacokinetic Pilot followed by a Phase I/II, Blinded, Randomized, Controlled, Parallel Arm Trial to Evaluate the Safety, Tolerability and Efficacy of PerioSept® and Scaling and Root Planing in Subjects with Periodontitis

DETAILED DESCRIPTION:
This trial will follow an adaptive trial design, whereby information regarding PerioSept(r) drug levels will be obtained via a PK trial lead in period (PK Pilot) in a limited number of subjects (up to N=8). This will be followed by the main safety and efficacy trial of PerioSept(r) as an adjunct to scaling and root planing (SRP) in subjects with moderate to severe periodontitis (Main Trial, N=87). The PK Pilot will be an open label PK study. Up to 8 qualifying subjects will receive SRP on Day 1 followed by 3% PerioSept(r) administered in a minimum of 4 qualifying periodontal Study Pockets in at least 2 quadrants with a probing pocket depth (PPD) ≥ 5mm and bleeding on probing (BOP) and at least 20 other qualifying pockets (PPD ≥ 5 mm). The Main Trial will be a multi-center, randomized, blinded, placebo controlled, parallel arm trial of PerioSept(r) (0.3%, 1% or 3%) administered up to three times (over Days 1 and 2, at Weeks 4 and 12) into a minimum of 4 qualifying periodontal Study Pockets in at least 2 quadrants with a PPD ≥ 5mm and BOP following SRP at baseline. All other eligible pockets with a PPD ≥ 5mm will also be treated.

Full mouth SRP will be initiated on Day 1 followed by randomized treatment of that side. If necessary, SRP and randomized treatment may be completed on the other side of the mouth on Day 2. Treated pockets that still have a PPD ≥ 5mm at the 4 and 12 week visits will be retreated with SRP or SRP plus placebo or PS, as randomized. Assessments will be conducted over a 24 week (6 month) period including safety assessments and assessments of dental parameters (PPD, BOP, Plaque index, Gingival Index, Clinical attachment level).

ELIGIBILITY:
Inclusion Criteria:

* 18 to 74 years of age, inclusive
* Diagnosed with moderate to severe generalized periodontitis (ADA Classification Case Type III or IV)
* Must have at least 4 qualifying Study Pockets (PPD ≥ 5mm and BOP) in at least 2 quadrants (main trial)
* Subjects must sign informed consent document(s) prior to initiation of any study-specific procedures and treatments
* Agree to utilize study-provided tooth paste and tooth brush and agree to follow their standard oral hygiene routine with limitations noted below from the Day 1 visit through the end of the study
* Sexually active subjects (both men and women) who agree to use acceptable contraceptive methods for the duration of the study
* Able and willing to adhere to the study visit schedule and other protocol requirements

Exclusion Criteria:

* History of and/or known risk of life-threatening anaphylactic reactions to taurolidine, any of the components in the PS drug product, and other drugs or agonists (e.g., penicillin, nuts, insect stings)
* Presence of an acute periodontal abscess
* Known endodontic disease
* Diabetes uncontrolled by medication defined as fasting blood glucose documented at ≥200 mg/dL within 90 days of Day 1
* History of illegal drug or alcohol abuse within the past 12 months and/or testing positive for illegal drugs (including marijuana) at the Screening Visit
* Pregnant or nursing female subjects; women of child-bearing potential must have a negative serum or urine pregnancy test within 30 days and within 24 h prior to all treatment/dosing days
* Use of systemic antibiotics and topically applied oral antibiotics and other antimicrobial agents (e.g., chlorhexidine) during the trial and within 30 days of Day 1.
* An existing condition that may warrant use of antibiotics during the trial (e.g., white blood cell count indicative of ongoing infection noted at Screening Visit, subject with cystic fibrosis or chronic obstructive pulmonary disorder with history of frequent, recurrent lung infections)
* History of and/or testing positive for Hepatitis B or C, Human Immunodeficiency Virus or other immunedeficiency syndrome or positive test for such at Screening Visit
* Use of chewing gum of any kind and dental flossing for one week after all study treatments and use of any other oral dentifrices or oral health agents/treatments other than those provided herein for the study duration
* Use within 30 days prior to Day 1, during trial or a condition for which use is anticipated during trial: topical oral, nasal and systemic corticosteroids, chronic (2 continuous weeks) non-steroidal anti-inflammatory drugs (NSAIDs)
* Use of the agents known to affect periodontal status during the trial and/or use within 30 days prior to Day 1: immunesuppressants, calcium antagonist, phenytoin or anticoagulants
* Heavy smokers/tobacco users are excluded: defined as those smoking ≥ 10 cigarettes or ≥ 4 cigars or ≥ 4 pipes per day
* For non-heavy smokers, smoking ≥ 10 cigarettes or ≥ 4 cigars or ≥ 4 pipes per day is prohibited for the duration of the trial
* Use of electronic/smokeless and herbal cigarettes/pipes and oral smokeless/chewing tobacco within 30 days of Day 1 excluded and all use of these products is prohibited during trial
* Clinically significant (e.g., QTc interval >450 milliseconds) abnormal electrocardiogram (ECG) noted at Screening Visit
* Participation in another clinical study with an investigational agent within 90 days prior to Day 1
* Subjects who received oral health treatments/interventions within 90 days of Day 1, which the investigator believes may interfere with the periodontal parameters to be assessed in this study (e.g., significant dental and/or gum/oral tissue work).
* Subject has a medical and/or dental condition and/or uses medications/supplements which the investigator believes makes him/her unsuitable for participation in the study

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2018-07-02 (Actual); Study Completion 2018-07-02 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability:Hematology safety labs, Chem 14, urine analysis, ECG, treatment emergent adverse events, local irritation, patient reported pain, sensisitivity, burning stinging | 6 months
  Hematology safety labs, Chem 14, urine analysis, ECG, treatment emergent adverse events, local irritation, patient reported pain, sensisitivity, burning stinging
Efficacy: Reduction in probing pocket depth (PPD) | 6 months
  Reduction in probing pocket depth (PPD)

SECONDARY OUTCOMES:
Efficacy REC and CAL: Changes from baseline in Recession (REC)/Clinical attachment level (CAL) | 6 months
  Changes from baseline in Recession (REC)/Clinical attachment level (CAL)
Efficacy BOP: Presence or absence of bleeding on probing (BOP) | 6 months
  Presence or absence of bleeding on probing (BOP)
Efficacy PI: Changes from baseline in Plaque index | 6 months
  Changes from baseline in Plaque index
Efficacy GI: Changes from baseline in Gingival index | 6 months
  Changes from baseline in Gingival index

OTHER OUTCOMES:
Efficacy microbial: Microbial Counts of Periodontal Pathogens | 6 months
  Microbial Counts of Periodontal Pathogens

CONTACTS AND LOCATIONS:
Overall Officials: Michael McGuire, DDS, Principal Investigator — PerioHealth Clinic Houston; Donald Clem, DDS, Principal Investigator — Regenerative Solutions; Tae-Ju Oh, DDS, Principal Investigator — University of Michigan
Locations (4):
- United States (4):
  - Regenerative solutions, Fullerton, California
  - University of Michigan School of Dentistry, Ann Arbor, Michigan
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Perio Health Professionals, Houston, Texas